CLINICAL TRIAL: NCT04388267
Title: Comparative Study on the Relationship Between Fluid REsponsiveness and Arterial ELASTANCE in Patients With Septic Shock or in the Postoperative Course of Aortic Surgery
Brief Title: Fluid REsponsiveness and Arterial ELASTANCE in Patients With Septic Shock or After Aortic Surgery
Acronym: RELASTANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/RELASTANCE-GUERCI/YB
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-01

CONDITIONS: Shock, Septic; Hyperlactatemia; Oliguria; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Ruptured; Aortic Stenosis
Keywords: Mostcare; Vascular surgery; Arterial Elastance; Dicrotic pressure; Fluid loading; Pressure Recording Analytical Method; Hemodynamic monitoring; Pulse contour analysis
MeSH Terms: conditions — Shock, Septic; Hyperlactatemia; Oliguria; Aortic Aneurysm, Abdominal; Aortic Rupture; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic shock: Patients with septic shock, according to the Sepsis 3 definition, regardless of the origin
  Interventions: Drug: Fluid challenge
- Major vascular surgery: Patients who underwent elective or emergent major vascular surgery abdominal aortic surgery (open or endovascular surgery)
  Interventions: Drug: Fluid challenge

INTERVENTIONS:
Drug: Fluid challenge — All patients who met the inclusion criteria will receive a standardised bolus of 250 ml of crystalloid in 5 minutes administered by hand with a 50 ml syringe.
  During the study period, hemodynamic parameters and analysis by pressure recording analytical method obtained with the MostCare will be collected for 20 minutes prior to the intervention (fluid challenge), during the fluid challenge and 25 minutes after completion.
  The total duration of the intervention (fluid loading) is 5 min. The total duration of hemodynamic parameters recording is 60 min.

SUMMARY:
The MostCare system, thanks to the Pressure Recording Analytical Method (PRAM; Vygon, Padua, Italy), provides new hemodynamic parameters of the cardiovascular system. The PRAM method is a noncalibrated pulse contour method which requires only an arterial line (radial or femoral). This method has been validated in various clinical conditions. Among the collected parameters, some are well known and used daily care in Intensive Care Unit (ICU), i.e. cardiac output (CO), arterial pressure, heart rate, stroke volume (SV). Others such as arterial elastance (Ea) or dicrotic pressure are more recent and merit further investigation to determine their interest in clinical practice. To date, it is rarely used to adapt therapies, mostly because of a lack of knowledge regarding the evolution of these parameters.

The aim of this study is to analyze the relationship between the evolution of Arterial Elastance and fluid responsiveness after a 250 mL fluid challenge of crystalloids in 5 minutes in patients with either septic shock or in the postoperative course of a major vascular surgery.

Patients will be considered fluid responders if an increase >10% of the stroke volume is observed .

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Septic shock (according to Sepsis-3 definition) or patients who underwent elective or emergent abdominal aortic surgery
* Invasive blood pressure (radial or femoral) and Mostcare monitoring
* Stroke volume between 20 and 50 mL/beat on the Mostcare system
* Indication for a fluid challenge: hypotension (Mean arterial pressure under 65mmHg) or oliguria (urine flow rate < 0,5mL/kg/h for more than 12h), mottling, hyperlactatemia > 2 mmol/l

Exclusion Criteria:

* Age <18 years
* Cardiac arrhythmia
* Arterial wave form distortion
* Inappropriate identification of the dicrotic notch for any reason
* Refuse to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a mix of septic shock and patients who underwent elective or emergent major vascular surgery surgery (aortic mostly) requiring a fluid challenge because of hypotension and/or oliguria and/or mottling and/or hyperlactatemia>2mmol/L. All patients will be hospitalized in the surgical intensive care unit (ICU) of the University Hospital of Nancy Brabois, France.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of arterial elastance | 60 minutes
  Absolute and percentage of change in arterial elastance during the study period
Evolution of Stroke Volume (SV) | 60 minutes
  Absolute and percentage of change in stroke volume during the study period

SECONDARY OUTCOMES:
Evolution of Dicrotic Pressure (DP) value during a fluid challenge | 60 minutes
  Absolute and percentage of change in dicrotic pressure during the study period
Predictive factors of an increase or a decrease in the arterial elastance value | 60 minutes
  Identification of clinical or arterial pressure waveform parameters associated with an increase or a decrease of the arterial elastance
  * epidemiological and clinical: age, BMI, gender, SAPS II, SOFA, Charlson comorbidity index, chronic diseases, etiology of the septic shock, acute kidney injury
  * therapeutical: chronic treatments, vasoactive and sedative drugs, epidural analgesia, mechanical ventilation (VT, RR, PEEP)
  * surgery: type of surgery (open or endovascular), indication, timing.
  * indication for fluid loading: hypotension, oliguria, hyperlactatemia > 2mmol/L, mottling
Predictive factors of an increase or a decrease of the dicrotic pressure value | 60 minutes
  Identification of clinical or arterial pressure waveform parameters associated with an increase or a decrease of the dicrotic pressure
Evolution of norepinephrine dose: before and 60 minutes after fluid challenge | 60 minutes
  Norepinephrine dose expressed in micrograms per kilogram per minute (μg/kg/min)
All-cause mortality | 30 days
  30 days all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Guerci, MD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU, Nancy, France

REFERENCES:
- [Background] Romagnoli S, Franchi F, Ricci Z, Scolletta S, Payen D. The Pressure Recording Analytical Method (PRAM): Technical Concepts and Literature Review. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1460-1470. doi: 10.1053/j.jvca.2016.09.004. Epub 2016 Sep 14. No abstract available. PMID 28012725
- [Background] Romagnoli S, Ricci Z, Romano SM, Dimizio F, Bonicolini E, Quattrone D, De Gaudio R. FloTrac/Vigileo(TM) (third generation) and MostCare((R))/PRAM versus echocardiography for cardiac output estimation in vascular surgery. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1114-21. doi: 10.1053/j.jvca.2013.04.017. Epub 2013 Sep 19. PMID 24055563
- [Background] Gopal S, Do T, Pooni JS, Martinelli G. Validation of cardiac output studies from the Mostcare compared to a pulmonary artery catheter in septic patients. Minerva Anestesiol. 2014 Mar;80(3):314-23. Epub 2014 Jan 8. PMID 24398442
- [Background] Messina A, Romano SM, Bonicolini E, Colombo D, Cammarota G, Chiostri M, Della Corte F, Navalesi P, Payen D, Romagnoli S. Cardiac cycle efficiency and dicrotic pressure variations: new parameters for fluid therapy: An observational study. Eur J Anaesthesiol. 2017 Nov;34(11):755-763. doi: 10.1097/EJA.0000000000000661. PMID 28722695
- [Background] Monge Garcia MI, Guijo Gonzalez P, Gracia Romero M, Gil Cano A, Oscier C, Rhodes A, Grounds RM, Cecconi M. Effects of fluid administration on arterial load in septic shock patients. Intensive Care Med. 2015 Jul;41(7):1247-55. doi: 10.1007/s00134-015-3898-7. Epub 2015 Jun 11. PMID 26077088
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Chantler PD, Lakatta EG, Najjar SS. Arterial-ventricular coupling: mechanistic insights into cardiovascular performance at rest and during exercise. J Appl Physiol (1985). 2008 Oct;105(4):1342-51. doi: 10.1152/japplphysiol.90600.2008. Epub 2008 Jul 10. PMID 18617626
- [Background] Sunagawa K, Maughan WL, Burkhoff D, Sagawa K. Left ventricular interaction with arterial load studied in isolated canine ventricle. Am J Physiol. 1983 Nov;245(5 Pt 1):H773-80. doi: 10.1152/ajpheart.1983.245.5.H773. PMID 6638199
- [Background] Guarracino F, Baldassarri R, Pinsky MR. Ventriculo-arterial decoupling in acutely altered hemodynamic states. Crit Care. 2013 Mar 19;17(2):213. doi: 10.1186/cc12522. No abstract available. PMID 23510336
- [Background] Suga H. Time course of left ventricular pressure-volume relationship under various enddiastolic volume. Jpn Heart J. 1969 Nov;10(6):509-15. doi: 10.1536/ihj.10.509. No abstract available. PMID 5308142
- [Background] Guarracino F, Ferro B, Morelli A, Bertini P, Baldassarri R, Pinsky MR. Ventriculoarterial decoupling in human septic shock. Crit Care. 2014 Apr 24;18(2):R80. doi: 10.1186/cc13842. PMID 24762124
- [Background] Morelli A, Singer M, Ranieri VM, D'Egidio A, Mascia L, Orecchioni A, Piscioneri F, Guarracino F, Greco E, Peruzzi M, Biondi-Zoccai G, Frati G, Romano SM. Heart rate reduction with esmolol is associated with improved arterial elastance in patients with septic shock: a prospective observational study. Intensive Care Med. 2016 Oct;42(10):1528-1534. doi: 10.1007/s00134-016-4351-2. Epub 2016 Apr 21. PMID 27101380
- [Background] Walley KR. Left ventricular function: time-varying elastance and left ventricular aortic coupling. Crit Care. 2016 Sep 10;20(1):270. doi: 10.1186/s13054-016-1439-6. PMID 27613430
- [Background] Guinot PG, Longrois D, Kamel S, Lorne E, Dupont H. Ventriculo-Arterial Coupling Analysis Predicts the Hemodynamic Response to Norepinephrine in Hypotensive Postoperative Patients: A Prospective Observational Study. Crit Care Med. 2018 Jan;46(1):e17-e25. doi: 10.1097/CCM.0000000000002772. PMID 29019850